CLINICAL TRIAL: NCT04620811
Title: A Phase 3, Multicenter, Open-Label, Extension Study to Evaluate the Efficacy and Safety of AK002 in Patients That Were Previously Enrolled in AK002-016 or AK002-012 Studies and Have Eosinophilic Gastritis and/or Eosinophilic Duodenitis (Formerly Referred to as Eosinophilic Gastroenteritis)
Brief Title: An Extension Study of Lirentelimab in Eosinophilic Gastritis and/or Eosinophilic Duodenitis (Formerly Referred to as Eosinophilic Gastroenteritis)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK002-016X
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Eosinophilic Gastritis; Eosinophilic Duodenitis
MeSH Terms: conditions — Eosinophilic enteropathy | interventions — AK002

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 3.0 mg/kg of Lirentelimab (AK002) (Experimental): Subjects in this arm will receive up to 18 monthly doses (3mg/kg) of lirentelimab (AK002)
  Interventions: Drug: lirentelimab

INTERVENTIONS:
Drug: lirentelimab — Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8
  Other Names: AK002

SUMMARY:
This is a Phase 3, open-label, extension study to assess the long term efficacy and safety of lirentelimab given monthly.

ELIGIBILITY:
Key Inclusion Criteria:

1. Provide written informed consent.
2. Completed Study AK002-016, defined as having received 6 infusions of study drug and followed through Day 176 (±3) or completed Study AK002-012, defined as having received the cohort-appropriate amount of doses and followed for 5 months after last dose of study drug.
3. If patient is on pre-existing dietary restrictions, willingness to maintain those restrictions, throughout the study.
4. Able and willing to comply with all study procedures.
5. Female patients must be either post-menopausal for at least 1 year or surgically sterile (tubal ligation, hysterectomy, or bilateral oophorectomy) for at least 3 months, or if of childbearing potential, have a negative pregnancy test and agree to use dual methods of contraception, or abstain from sexual activity until the end of the study, or for 120 days following the last dose of study drug, whichever is longer.
6. Male patients with female partners of childbearing potential must agree to use a highly effective method of contraception until the end of the study or for 120 days following the last dose of study drug, whichever is longer. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant at any time during study participation.

Key Exclusion Criteria:

1. Known hypersensitivity to any constituent of the study drug.
2. Any disease, condition (medical or surgical), or cardiac abnormality, which, in the opinion of the Investigator, would place the patient at increased risk.
3. Planned or expected vaccination with live attenuated vaccines during the Treatment Period, or vaccination expected within 5 half-lives (4 months) of AK002 administration.
4. Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study.
5. Any other reason that, in the opinion of the Investigator or Medical Monitor, makes the patient unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Patterson, MD, Study Director — Allakos Inc.
Locations (38):
- United States (38):
  - Allakos Investigational Site 216-068, Birmingham, Alabama
  - Allakos Investigational Site 216-002, Huntsville, Alabama
  - Allakos Investigational Site 216-035, Phoenix, Arizona
  - Allakos Investigational Site 216-032, Chula Vista, California
  - Allakos Investigational Site 216-014, Santa Monica, California
  - Allakos Investigational Site 216-038, Tustin, California
  - Allakos Investigational Site 216-049, Walnut Creek, California
  - Allakos Investigational Site 216-034, Aurora, Colorado
  - Allakos Investigational Site 216-063, Brandon, Florida
  - Allakos Investigational Site 216-027, Edgewater, Florida
  - Allakos Investigational Site 216-056, Jacksonville, Florida
  - Allakos Investigational Site 216-013, Miami, Florida
  - Allakos Investigational Site 216-053, New Port Richey, Florida
  - Allakos Investigational Site 216-007, Chicago, Illinois
  - Allakos Investigational Site 216-001, Crowley, Louisiana
  - Allakos Investigational Site 216-026, Boston, Massachusetts
  - Allakos Investigational Site 216-052, Boston, Massachusetts
  - Allakos Investigational Site 216-051, Boston, Massachusetts
  - Allakos Investigational Site 216-005, Rochester, Minnesota
  - Allakos Investigational Site 216-042, Kansas City, Missouri
  - Allakos Investigational Site 216-045, Reno, Nevada
  - Allakos Investigational Site 216-025, New York, New York
  - Allakos Investigational Site 216-020, Chapel Hill, North Carolina
  - Allakos Investigational Site 216-048, Durham, North Carolina
  - Allakos Investigational Site 216-050, Winston-Salem, North Carolina
  - Allakos Investigational Site 216-031, Cincinnati, Ohio
  - Allakos Investigational Site 216-028, Cincinnati, Ohio
  - Allakos Investigational Site 216-044, Mentor, Ohio
  - Allakos Investigational Site 216-021, Philadelphia, Pennsylvania
  - Allakos Investigational Site 216-006, Chattanooga, Tennessee
  - Allakos Investigational Site 216-003, Chattanooga, Tennessee
  - Allakos Investigational Site 216-011, Chattanooga, Tennessee
  - Allakos Investigational Site 216-062, Kingsport, Tennessee
  - Allakos Investigational Site 216-022, Austin, Texas
  - Allakos Investigational Site 216-039, Ogden, Utah
  - Allakos Investigational Site 216-030, Salt Lake City, Utah
  - Allakos Investigational Site 216-055, Sandy City, Utah
  - Allakos Investigational Site 216-064, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants who were enrolled in and completed the studies AK002-016 (NCT04322604) or AK002-012 had the option to participate in this open-label extension study.
Groups:
- Main Study Placebo to Extension Study 3.0 mg/kg of Lirentelimab (AK002): Subjects in this arm received the placebo in the main study and were treated with up to 18 monthly doses (3mg/kg) of lirentelimab (AK002).
  lirentelimab: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8.
- Main Study Active to Extension Study 3.0 mg/kg of Lirentelimab (AK002): Subjects in this arm received the active drug in the main study and were treated with up to 18 monthly doses (3mg/kg) of lirentelimab (AK002).
  lirentelimab: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8.
Period: Overall Study
Arm/Group | Main Study Placebo to Extension Study 3.0 mg/kg of Lirentelimab (AK002) | Main Study Active to Extension Study 3.0 mg/kg of Lirentelimab (AK002)
Started | 75 | 84
Completed | 42 | 40
Not Completed | 33 | 44
Not completed — Withdrawal by Subject | 18 | 15
Not completed — Adverse Event | 6 | 11
Not completed — Lost to Follow-up | 4 | 8
Not completed — Physician Decision | 1 | 4
Not completed — Sponsor Decision | 0 | 1
Not completed — Elevation of ALT or AST | 1 | 0
Not completed — Other | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study Placebo to Extension Study 3.0 mg/kg of Lirentelimab (AK002) | Main Study Active to Extension Study 3.0 mg/kg of Lirentelimab (AK002) | Total
Number analyzed (Participants) | 75 | 84 | 159
Age, Continuous [Median (Full Range); unit: years] | 42 [18 to 79] | 42 [18 to 77] | 42 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 53 | 103
  Male | 25 | 31 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 13 | 23
  Not Hispanic or Latino | 65 | 71 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 5 | 7 | 12
  White | 66 | 68 | 134
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75 | 84 | 159

OUTCOME MEASURES:

1. Primary Outcome: The Safety and Tolerability of Lirentelimab by Evaluating Adverse Events Assessed Using the CTCAE Version 5.0
Description: Adverse events assessed using the CTCAE version 5.0.
Time Frame: Through study completion, up to 21 months
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Placebo to Extension Study 3.0 mg/kg of Lirentelimab (AK002) | Main Study Active to Extension Study 3.0 mg/kg of Lirentelimab (AK002)
Number analyzed (Participants) | 75 | 84
Participants
  No. of Subjects with >=1 Adverse Events | 66 | 75
  No. of Subjects with >=1 Treatment-Related Adverse Events | 33 | 29
  No. of Subjects with >=1 Serious Adverse Events | 6 | 14
  No. of Subjects with an Adverse Event Leading to Study Drug Discontinuation | 6 | 10
  No. of Subjects with >=1 Treatment-Related Serious Adverse Events | 1 | 1

2. Other Pre Specified Outcome: Proportion of Tissue Eosinophil Responders
Description: A tissue eosinophil responder is defined as mean eosinophil count ≤4 cells/HPF in 5 gastric HPFs for EG only patients, ≤15 cells/HPF in 3 duodenal HPFs for EoD only patients, and ≤4 cells/HPF in 5 gastric HPFs and ≤15 cells/HPF in 3 duodenal HPFs for EG+EoD patients.
Time Frame: At Follow-up EGD (Esophago-Gastro-Duodenoscopy) (Day 505 or 28 days after last dose if ET)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Placebo to Extension Study 3.0 mg/kg of Lirentelimab (AK002) | Main Study Active to Extension Study 3.0 mg/kg of Lirentelimab (AK002)
Number analyzed (Participants) | 54 | 52
Participants | 52 | 48

3. Other Pre Specified Outcome: Change in PRO Total System Score (TSS) From AK002-016/AK002-012 Baseline
Description: The PRO Total Symptom Score (TSS) is a patient reported outcome (PRO) questionnaire comprises the following 6 symptoms: Abdominal pain intensity, Nausea intensity, Fullness before meal intensity, Loss of appetite intensity, Bloating intensity, and Abdominal cramping intensity. TSS scores can range from 0 to 60, with a lower score indicating less-severe symptoms.
Time Frame: Main Study Baseline to Extension Weeks 71-72
Population: Number of participants with available data within Safety Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main Study Placebo to Extension Study 3.0 mg/kg of Lirentelimab (AK002) | Main Study Active to Extension Study 3.0 mg/kg of Lirentelimab (AK002)
Number analyzed (Participants) | 46 | 41
score on a scale | -14.4 (11.0) | -17.0 (12.1)

ADVERSE EVENTS:
Time Frame: Through study completion, up to 21 months
Description: NCI Common Terminology Criteria for Adverse Events Version (CTCAE) 5.0 or most current version
Arm/Group | Main Study Placebo to Extension Study 3.0 mg/kg of Lirentelimab (AK002) | Main Study Active to Extension Study 3.0 mg/kg of Lirentelimab (AK002)
All-Cause Mortality (participants affected / at risk) | 0/75 | 1/84
Serious Adverse Events (participants affected / at risk) | 6/75 | 14/84
Other Adverse Events (participants affected / at risk) | 52/75 | 57/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study Placebo to Extension Study 3.0 mg/kg of Lirentelimab (AK002) (N=75) | Main Study Active to Extension Study 3.0 mg/kg of Lirentelimab (AK002) (N=84)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 2 | 0
Meningitis viral (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Radial nerve palsy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aortic thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study Placebo to Extension Study 3.0 mg/kg of Lirentelimab (AK002) (N=75) | Main Study Active to Extension Study 3.0 mg/kg of Lirentelimab (AK002) (N=84)
Anaemia (Blood and lymphatic system disorders) | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 7 | 9
Diarrhoea (Gastrointestinal disorders) | 11 | 8
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 11 | 5
Vomiting (Gastrointestinal disorders) | 3 | 10
Hypersensitivity (Immune system disorders) | 4 | 2
Corona virus infection (Infections and infestations) | 15 | 21
Nasopharyngitis (Infections and infestations) | 6 | 4
Sinusitis (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 8 | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 27 | 19
Coronavirus test positive (Investigations) | 1 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Headache (Nervous system disorders) | 6 | 7
Depression (Psychiatric disorders) | 0 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement contains a limit on publication of results following completion of the trial. PIs are not allowed to publish results until a joint publication for the multicenter study or a set period of time. After that time, PIs may only publish results from their portion of the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT04620811/Prot_SAP_000.pdf